CLINICAL TRIAL: NCT01475825
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Followed by an Open-Label Continuation Period to Assess the Safety and Efficacy of Two Different Regimens of Mipomersen in Patients With Familial Hypercholesterolemia and Inadequately Controlled Low-Density Lipoprotein Cholesterol
Brief Title: A Study of the Safety and Efficacy of Two Different Regimens of Mipomersen in Patients With Familial Hypercholesterolemia and Inadequately Controlled Low-Density Lipoprotein Cholesterol
Acronym: FOCUS FH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIPO3801011; 2011-001480-42 (EudraCT Number); EFC12875 (Other: Sanofi)
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Hypercholesterolemia; Heterozygous Familial
MeSH Terms: conditions — Hypercholesterolemia | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen A: Mipomersen (Experimental): Subcutaneous injection of mipomersen 200 mg once weekly
  Interventions: Drug: mipomersen sodium 200 mg
- Regimen A: Placebo (Placebo Comparator): Placebo matching subcutaneous injection once weekly.
  Interventions: Drug: Placebo
- Regimen B: Mipomersen (Experimental): Subcutaneous injection of mipomersen 70 mg thrice weekly.
  Interventions: Drug: mipomersen sodium 70 mg
- Regimen B: Placebo (Placebo Comparator): Placebo matching subcutaneous injection thrice weekly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mipomersen sodium 200 mg — Subcutaneous mipomersen 200 mg once weekly
  Other Names: Kynamro (ISIS 301012)
  Arms: Regimen A: Mipomersen
Drug: Placebo — Placebo vehicle for subcutaneous injection.
  Arms: Regimen A: Placebo; Regimen B: Placebo
Drug: mipomersen sodium 70 mg — Subcutaneous mipomersen 70 mg thrice weekly
  Other Names: Kynamro (ISIS 301012)
  Arms: Regimen B: Mipomersen

SUMMARY:
Primary objective:

Determine whether mipomersen (ISIS 301012) significantly reduces atherogenic lipid levels in patients with severe heterozygous familial hypercholesterolemia (severe HeFH), defined as low-density lipoprotein cholesterol (LDL-C) levels ≥200 mg/dL plus the presence of coronary heart disease (CHD)/risk equivalents or LDL-C levels ≥300 mg/dL regardless of the presence of CHD/risk equivalents (referred to as Cohort 1) compared to placebo. Two different mipomersen dosing regimens will be studied: subcutaneous (SC) mipomersen 200 mg once weekly versus placebo, and SC mipomersen 70 mg thrice weekly versus placebo.

Secondary Objectives:

* Determine whether there are qualitative differences between the safety profiles of the 2 dosing regimens and placebo in Cohort 1, patients with HeFH with LDL-C levels ≥160 mg/dL and <200 mg/dL plus the presence of CHD/risk equivalents (referred to as Cohort 2), and the overall study population
* Determine whether there are qualitative differences between the tolerability of the 2 dosing regimens and placebo in Cohort 1, Cohort 2, and the overall study population
* Further characterize the pharmacokinetics (PK) of the 2 dosing regimens in Cohort 1, Cohort 2, and the overall study population
* Determine whether the 2 mipomersen dosing regimens significantly reduce atherogenic lipid levels in Cohort 2 compared to placebo
* Obtain additional data regarding ongoing safety and efficacy of mipomersen in patients with FH and inadequately controlled LDL-C who complete the primary efficacy assessment visit (PET) in the Blinded Treatment Period and continue treatment in Open-Label Continuation Period

DETAILED DESCRIPTION:
The study consisted of a Screening period of up to 4 weeks, Blinded Treatment Phase of 60 weeks, Open-Label Continuation Period of 26 weeks, and Post-Treatment Phase of 24 weeks.

Study Design, masking - Study treatment was blinded (double-blinded) through the Primary Efficacy Assessment Visit in the Blinded Treatment Period. Study treatment was open-label in the Open-Label Continuation Period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe hypercholesterolemia (LDL-C ≥300 mg/dL (7.77 mmol/L) or LDL-C ≥200 mg/dL (5.18 mmol/L) with documented coronary heart disease (CHD) or CHD risk equivalents, or diagnosis of Heterozygous Familial Hypercholesterolemia and LDL-C ≥160 mg/dL (4.14 mmol/L) and <200 mg/dL (5.18 mmol/L))
* On stable, maximally tolerated, statin therapy for at least 12 weeks or if statin intolerant, on at least 1 medication from another class of hypolipidemic agents (i.e., bile acid sequestrants, niacin/nicotinic acid, cholesterol absorption inhibitors, fibrates).
* On stable, low fat diet for 12 weeks
* Body mass index (BMI) ≤40 kg/m2 and stable weight for > 6 weeks

Exclusion Criteria:

* Significant health problems in the recent past including heart attack, stroke, coronary syndrome, unstable angina, heart failure, significant arrhythmia, hypertension, blood disorders, liver disease, cancer, digestive disorders, Type I diabetes, or uncontrolled Type II diabetes
* Apheresis within 3 months prior to Screening or expected to start apheresis during the treatment phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2015-12-29 (Actual); Study Completion 2015-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (113):
- United States (20):
  - Mission Viejo, California
  - Aurora, Colorado
  - Cooper City, Florida
  - Winter Park, Florida
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Grandville, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Summit, New Jersey
  - North Massapequa, New York
  - Portland, Oregon
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Norfolk, Virginia
- Argentina (2):
  - Buenos Aires
  - Córdoba
- Australia (2):
  - Perth
  - South Brisbane
- Belgium (3):
  - Edegem
  - Haine-Saint-Paul
  - Leuven
- Brazil (2):
  - Rio de Janeiro
  - São Paulo
- Canada (3):
  - Chicoutimi, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec
- Croatia (2):
  - Osijek
  - Zagreb
- Czechia (2):
  - Hradec Králové
  - Prague
- Denmark (2):
  - Aarhus
  - Viborg
- Germany (7):
  - Aachen
  - Berlin
  - Cologne
  - Freiburg im Breisgau
  - Hamburg
  - Heidelberg
  - Magdeburg
- Greece (2):
  - Ioannina
  - Kallithea
- Hong Kong, Hong Kong
- Hungary (3):
  - Baja
  - Budapest
  - Debrecen
- New Delhi, India
- Israel (3):
  - Holon
  - Kfar Saba
  - Ofakim
- Italy (6):
  - Bologna
  - Napoli
  - Padua
  - Palermo
  - Pisa
  - Roma
- Malaysia (2):
  - Kuala Lumpur
  - Kubang Kerian
- Netherlands (6):
  - Alkmaar
  - Amsterdam
  - Maastricht
  - Nijmegen
  - Utrecht
  - Waalwijk
- Christchurch, New Zealand
- Norway (3):
  - Bodø
  - Oslo
  - Sandefjord
- Poland (10):
  - Bialystok
  - Gdansk
  - Katowice
  - Krakow
  - Nałęczów
  - Poznan
  - Sopot
  - Szczecin
  - Warsaw
  - Wroclaw
- Russia (9):
  - Barnaul
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Ryazan
  - Saint Petersburg
  - Tomsk
  - Yaroslavl
- South Africa (2):
  - Cape Town
  - Pretoria
- Seoul, South Korea
- Madrid, Spain
- Stockholm, Sweden
- Taiwan (2):
  - New Taipei City
  - Taipei
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Sivas
- Ukraine (4):
  - Ivano-Frankivsk
  - Kiev
  - Kyiv
  - Odesa
- United Kingdom (6):
  - Birmingham
  - Cardiff
  - Liverpool
  - London
  - Manchester
  - Oldham

REFERENCES:
- [Derived] Tragante V, Asselbergs FW, Swerdlow DI, Palmer TM, Moore JH, de Bakker PIW, Keating BJ, Holmes MV. Harnessing publicly available genetic data to prioritize lipid modifying therapeutic targets for prevention of coronary heart disease based on dysglycemic risk. Hum Genet. 2016 May;135(5):453-467. doi: 10.1007/s00439-016-1647-9. Epub 2016 Mar 5. PMID 26946290

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: Mipomersen, 200 mg, Once Weekly: Participants received once weekly subcutaneous (SC) injections of mipomersen sodium 200 milligrams (mg) during the 60-week Blinded Treatment Period, continued the dosing regimen during the 26-week Open-Label Continuation Period, and then entered the 24-week Post-Treatment Period.
- Regimen A: Placebo, Once Weekly: Participants received once weekly SC injections of Placebo during the 60-week Blinded Treatment Period, continued the dosing regimen during the 26-week Open-Label Continuation Period, and then entered the 24-week Post-Treatment Period.
- Regimen B: Mipomersen, 70 mg, Thrice Weekly: Participants received thrice weekly SC injections of mipomersen sodium 70 mg during the 60-week Blinded Treatment Period, continued the dosing regimen during the 26-week Open-Label Continuation Period, and then entered the 24-week Post-Treatment Period.
- Regimen B: Placebo, Thrice Weekly: Participants received thrice weekly SC injections of placebo during the 60-week Blinded Treatment Period, continued the dosing regimen during the 26-week Open-Label Continuation Period, and then entered the 24-week Post-Treatment Period.
Period: Overall Study
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Started | 104 | 51 | 102 | 52
Randomized and Treated | 104 | 51 | 102 | 52
Completed Blinded Treatment Period | 60 | 42 | 59 | 40
Entered Open-Label Continuation | 45 | 31 | 44 | 29
Completed Open-Label Continuation | 37 | 19 | 38 | 22
Completed | 37 | 19 | 38 | 22
Not Completed | 67 | 32 | 64 | 30
Not completed — Adverse Event | 41 | 15 | 27 | 11
Not completed — Death | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Non-compliance with Study Drug | 1 | 2 | 4 | 0
Not completed — Other: Not available | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 3 | 11 | 7
Not completed — Did not enter OLC | 15 | 11 | 15 | 11

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who took at least 1 dose of study drug (mipomersen or placebo), had a valid baseline low-density lipoprotein cholesterol (LDL-C) measurement, and had at least 1 post-baseline LDL-C measurement.
Groups:
- Regimen A: Mipomersen, 200 mg, Once Weekly: Participants received once weekly SC injections of mipomersen sodium 200 mg during the 60-week Blinded Treatment Period, continued the dosing regimen during the 26-week Open-Label Continuation Period, and then entered the 24-week Post-Treatment Period.
- Total: Total of all reporting groups
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly | Total
Number analyzed (Participants) | 104 | 51 | 102 | 52 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.36 (9.766) | 55.49 (10.481) | 53.15 (11.918) | 54.38 (9.939) | 54.85 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 29 | 54 | 27 | 168
  Male | 46 | 22 | 48 | 25 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 4 | 6 | 18
  Not Hispanic or Latino | 99 | 45 | 95 | 46 | 285
  Unknown or Not Reported | 1 | 2 | 3 | 0 | 6
LDL-C Baseline Values [Mean (Standard Deviation); unit: mg/dL] — Population: The full analysis set was analyzed in two cohorts, shown below.
  mg/dL
    Cohort 1: number analyzed (Participants) | 67 | 34 | 66 | 33 | 200
    Cohort 1 | 262 (103.1) | 255 (75.0) | 274 (75.1) | 263 (82.9) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis
    Cohort 2: number analyzed (Participants) | 37 | 17 | 36 | 19 | 109
    Cohort 2 | 177 (20.8) | 179 (25.6) | 178 (17.6) | 169 (26.6) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis
Apolipoprotein B Baseline Values [Mean (Standard Deviation); unit: mg/dL] — Population: The full analysis set was analyzed in two cohorts, shown below.
  mg/dL
    Cohort 1: number analyzed (Participants) | 67 | 34 | 66 | 33 | 200
    Cohort 1 | 172 (52.1) | 170 (35.0) | 182 (37.9) | 174 (45.2) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis
    Cohort 2: number analyzed (Participants) | 37 | 17 | 36 | 19 | 109
    Cohort 2 | 131 (17.3) | 134 (17.0) | 135 (16.3) | 128 (23.4) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis
Lipoprotein (a) Baseline Values [Mean (Standard Deviation); unit: mg/dL] — Population: The full analysis set was analyzed in two cohorts, shown below.
  mg/dL
    Cohort 1: number analyzed (Participants) | 67 | 34 | 66 | 33 | 200
    Cohort 1 | 43 (39.5) | 50 (45.6) | 38 (40.3) | 51 (50.8) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis
    Cohort 2: number analyzed (Participants) | 37 | 17 | 36 | 19 | 109
    Cohort 2 | 52 (58.4) | 48 (65.6) | 59 (49.3) | 27 (28.2) | NA (NA) — The total baseline values were not originally calculated, and data were no longer available for further analysis

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline To Primary Endpoint Visit (PET) In LDL-C In Cohort 1
Description: The percent change from baseline to PET in LDL-C was measured in Cohort 1, which included participants with severe heterozygous familial hypercholesterolemia (HeFH). Severe HeFH was defined as LDL-C levels ≥200 mg/deciliter (dL) plus the presence of coronary heart disease (CHD)/risk equivalents or LDL-C levels ≥300 mg/dL regardless of the presence of CHD/risk equivalents.
Time Frame: Baseline and Week 61
Population: The full analysis set for Cohort 1 included all randomized participants who took at least 1 dose of study drug in Cohort 1 (mipomersen or placebo), had a valid baseline LDL-C measurement, and had at least 1 post-baseline LDL-C measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 67 | 34 | 66 | 33
Percent | -27.17 (5.653) | -6.77 (6.749) | -22.96 (5.362) | -10.62 (5.765)

2. Secondary Outcome: Percent Change From Baseline To PET In LDL-C In Cohort 2
Description: The percent change from baseline to PET in LDL-C was measured in Cohort 2, which included participants with HeFH with LDL-C levels ≥160 mg/dL and <200 mg/dL, plus the presence of CHD/risk equivalents.
Time Frame: Baseline, PET (up to 60 weeks)
Population: The full analysis set included all randomized participants who took at least 1 dose of study drug (mipomersen or placebo), had a valid baseline LDL-C measurement, and had at least 1 post-baseline LDL-C measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 37 | 17 | 36 | 19
Percent | -31.20 (8.927) | -9.25 (10.621) | -43.60 (8.342) | -13.57 (9.066)

3. Secondary Outcome: Percent Change From Baseline To PET In Apolipoprotein B (Apo B) In Cohort 1
Description: The percent change from baseline to PET in Apo B was measured in participants in Cohort 1 with HeFH during the Blinded Treatment Period.
Time Frame: Baseline and Week 61
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 67 | 34 | 66 | 33
Percent | -24.14 (5.058) | -2.83 (6.115) | -21.43 (4.861) | -7.28 (5.309)

4. Secondary Outcome: Percent Change From Baseline To PET In Apolipoprotein B (Apo B) In Cohort 2
Description: The percent change from baseline to PET in Apo B was measured in participants in Cohort 2 with HeFH during the Blinded Treatment Period.
Time Frame: Baseline and Week 61
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 37 | 17 | 36 | 19
Percent | -30.76 (7.309) | -6.67 (8.758) | -36.34 (7.039) | -3.77 (8.109)

5. Secondary Outcome: Percent Change From Baseline To PET in Lipoprotein (a) In Cohort 1
Description: The percent change from baseline to PET in Lipoprotein A1 was measured in participants in Cohort 1 with HeFH during the Blinded Treatment Period.
Time Frame: Baseline and Week 61
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 67 | 34 | 66 | 33
Percent | -18.84 (7.870) | -16.85 (9.959) | -27.18 (5.497) | -10.08 (5.992)

6. Secondary Outcome: Percent Change From Baseline To PET in Lipoprotein (a) In Cohort 2
Description: The percent change from baseline to PET in Lipoprotein A1 was measured in participants in Cohort 2 with HeFH during the Blinded Treatment Period.
Time Frame: Baseline and Week 61
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
Number analyzed (Participants) | 37 | 17 | 36 | 19
Percent | -23.41 (10.002) | -11.86 (11.871) | -35.56 (11.846) | 18.79 (15.271)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of the administration of the participant's first dose of study drug (mipomersen or placebo) through the participant's last visit of the Post-Treatment Period, up to Week 110.
Description: Adverse events were collected for all randomized participants who received at least 1 dose of study drug (mipomersen or placebo).
Arm/Group | Regimen A: Mipomersen, 200 mg, Once Weekly | Regimen A: Placebo, Once Weekly | Regimen B: Mipomersen, 70 mg, Thrice Weekly | Regimen B: Placebo, Thrice Weekly
All-Cause Mortality (participants affected / at risk) | 1/104 | 0/51 | 1/102 | 0/52
Serious Adverse Events (participants affected / at risk) | 17/104 | 13/51 | 23/102 | 11/52
Other Adverse Events (participants affected / at risk) | 82/104 | 27/51 | 78/102 | 33/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Mipomersen, 200 mg, Once Weekly (N=104) | Regimen A: Placebo, Once Weekly (N=51) | Regimen B: Mipomersen, 70 mg, Thrice Weekly (N=102) | Regimen B: Placebo, Thrice Weekly (N=52)
Angina pectoris (Cardiac disorders) | 7 | 4 | 0 | 4
Angina unstable (Cardiac disorders) | 1 | 3 | 4 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 2 | 2
Coronary artery disease (Cardiac disorders) | 3 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 3 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 2 | 0
Death (General disorders) | 2 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Helicobacter test negative (Investigations) | 0 | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Mipomersen, 200 mg, Once Weekly (N=104) | Regimen A: Placebo, Once Weekly (N=51) | Regimen B: Mipomersen, 70 mg, Thrice Weekly (N=102) | Regimen B: Placebo, Thrice Weekly (N=52)
Influenza like illness (General disorders) | 43 | 10 | 26 | 10
Injection site erythema (General disorders) | 8 | 1 | 13 | 1
Injection site pain (General disorders) | 13 | 1 | 7 | 0
Injection site swelling (General disorders) | 4 | 1 | 8 | 1
Injection site pruritus (General disorders) | 3 | 1 | 7 | 1
Nasopharyngitis (Infections and infestations) | 7 | 4 | 7 | 7
Influenza (Infections and infestations) | 5 | 3 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 7 | 2
Bronchitis (Infections and infestations) | 5 | 3 | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 0 | 7 | 1
Alanine aminotransferase increased (Investigations) | 21 | 2 | 18 | 0
Aspartate aminotransferase increased (Investigations) | 17 | 2 | 11 | 1
C-reactive protein increased (Investigations) | 4 | 3 | 3 | 3
Hepatic enzyme increased (Investigations) | 8 | 0 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 0
Headache (Nervous system disorders) | 8 | 2 | 9 | 4
Dizziness (Nervous system disorders) | 8 | 1 | 3 | 1
Angina pectoris (Cardiac disorders) | 8 | 5 | 4 | 6
Palpitations (Cardiac disorders) | 2 | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 9 | 3 | 7 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 10 | 1 | 9 | 1
Hypertension (Vascular disorders) | 3 | 3 | 4 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days